CLINICAL TRIAL: NCT01485055
Title: Infliximab and Basiliximab for Treatment of Steroid Refractory Acute Graft Versus Host Disease
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor withdrew support
Sponsor: Nationwide Children's Hospital (Other)
Responsible Party: Principal Investigator, Rajinder Bajwa, Rajinder.P.S. Bajwa, MBBS, MD, MRCP Assitant Professor of Pediatrics at Ohio State University Department of Hematology/Oncology/BMT, Nationwide Children's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCH-IRB11-00659
Record Dates: First submitted 2011-12-01; First posted 2011-12-05 (Estimated); Results first posted 2019-04-05 (Actual); Last update posted 2019-04-05 (Actual); Status verified 2019-04

CONDITIONS: Graft Versus Host Disease; Steroid Refractory GVHD; Acute GVH Disease
Keywords: aGVHD; GVHD; Graft versus host disease; Acute graft versus host disease; Steroid refractory graft versus host disease; Bone marrow transplant; BMT; HSCT; infliximab; basiliximab; Monoclonal antibody treatment
MeSH Terms: conditions — Graft vs Host Disease | interventions — Infliximab; Basiliximab; Antibodies, Monoclonal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Infliximab and Basiliximab (Experimental): Other Names:
  Simulect Remicade Monoclonal antibody
  Participants in this research study will receive combination therapy (2 drugs: Infliximab and Basiliximab)once a week for four weeks. Both drugs will be given through the participant's broviac, port or through a vein in the arm. It will take about 4-5 hours to complete the 2-drug combination therapy each week. Participants will be given pre-medications to help prevent reactions to the study drugs.
  Infliximab will be given at a dose of 10mg per Kg per dose. Basiliximab will be given in 10mg doses to patients who weigh less than 35kg. Patients who weigh weigh more than 35kg will receive 20mg doses. Patients will receive both drugs weekly on days 1,8,15 and 22. Each drug will be given 4 times.
  Interventions: Drug: Infliximab and Basiliximab

INTERVENTIONS:
Drug: Infliximab and Basiliximab — Participants in this research study will receive combination therapy (2 drugs: Infliximab and Basiliximab)once a week for four weeks. Both drugs will be given through the participant's broviac, port or through a vein in the arm. It will take about 4-5 hours to complete the 2-drug combination therapy each week. Participants will be given pre-medications to help prevent reactions to the study drugs.
  Infliximab will be given at a dose of 10mg per Kg per dose. Basiliximab will be given in 10mg doses to patients who weigh less than 35kg. Patients who weigh weigh more than 35kg will receive 20mg doses. Patients will receive both drugs weekly on days 1,8,15 and 22. Each drug will be given 4 times.
  Other Names: Simulect; Remicade; Monoclonal antibody

SUMMARY:
Acute Graft Versus Host Disease (GVHD) is a serious medical condition that is a common development after Bone Marrow Transplant (BMT). Acute GVHD happens when the donor cells attack and damage your tissues and organs after transplant.

Acute GVHD often causes: Skin rashes, nausea, vomiting, abdominal pain, diarrhea (may have blood), liver damage that can cause inflammation in the liver or jaundice (yellowing of the skin or eyes), damage to other organs

Steroids are the first line of treatment for acute GVHD. About a quarter of the patients that develop acute GVHD may not respond to steroid and have steroid refractory GVHD (SR-aGVHD). Patients with SR-aGVHD may need other medications. SR-aGVHD, is a potentially life threatening condition. There is no standard treatment and it may not respond to treatment.

The goals of this study are to find out if Infliximab and basiliximab can treat SR-aGVHD.

Participants in this study will receive combination therapy (2 drugs: infliximab and basiliximab) once a week for four weeks.

DETAILED DESCRIPTION:
Corticosteroids are the standard initial therapy for Acute GvHD (aGVHD) after HSCT (hematopoietic stem cell transplant aka BMT) and 25-41% patients will respond to prednisone (or methylprednisolone) at a dose of 2mg/kg/day. Complete response of aGvHD is an important predictor of survival; in patients who respond to steroids, survival is around 50%, while it is as low as 11% for non-responders. Patients who do not develop aGvHD are normally discharged by 4-5 weeks after HSCT. However patients with aGvHD may need to be admitted and require prolonged hospitalization. Patients, who do not respond to treatment, usually have worsening skin symptoms, the protracted diarrhea and vomiting leading to severe life threatening dehydration. Secondary bacterial, fungal and/or viral infections are common and they may eventually die of multiorgan failure.

There is no consensus to the definition of steroid refractory (SR) aGvHD, but generally aGvHD is considered to be SR, when there is progression of GvHD after 3 days or no response after 7 days of treatment with 2mg/kg/day of methyl prednisolone. There is no standard of care for such patients and treatment varies from institution to institution. Salvage regimens for SR GvHD have included high dose steroids, antithymocyte globulin (ATG), monoclonal antibodies (infliximab, daclizumab, basiliximab etc.),pentostatin, mesenchymal stem cells and immunotoxins. Generally if the manifestations of aGvHD worsen over 3 days after starting steroids, or if there is no improvement within 5 days, then it is unlikely that a response will be achieved and secondary therapy should be initiated.

High dose steroids have not been associated with any improvement in response rates for SR aGvHD. In a prospective trial comparing 2mg/kg/day with 10mg/kg/day of methylprednisolone in 94 patients with grade II-IV aGvHD, response rates, progression to grade III-IV disease, non- relapse mortality (NRM) and overall survival were similar in both treatment groups. In addition high dose steroids are associated with many acute and long term complications. Hyperglycemia, hypertension, infections, aseptic necrosis and neurological complications are commonly seen.

Outcome of patients with SR aGvHD is poor. Only 7/57 (12%) patients achieved CR (complete Response)after secondary therapy for aGvHD as reported by Weisdorf et al and only 4/45 (9 %) patients who received high dose methylprednisolone as secondary therapy responded. ATG has been extensively used for treatment of SR GvHD and CR rates of 14-20 % have been reported.

Rationale for using Infliximab and Basiliximab:

The pathophysiology of GvHD is triphasic involving tissue damage from the conditioning regimen, followed by donor T cell activation leading to the effector phase of cytokine dysregulation. The cytokines interleukin (IL) 2 and tumor necrosis factor-α (TNF-α) play a central role in mediating tissue damage and causing proliferation of the activated alloreactive T cells. Over the last few years monoclonal antibodies have been used to treat such patients as monotherapy and recently as combination therapy with more promising results. The anti-CD25 MoAb - daclizumab provides competitive inhibition of binding of IL-2 to the high affinity α subunit IL2 receptor. It has been used as monotherapy for steroid refractory aGvHD with promising results. TNF is another cytokine involved in GvHD and early studies with anti-TNF-α administration have shown encouraging results. Antibodies to TNF (infliximab) or to TNF receptor (etanercept) have been developed. Infliximab blocks the interaction between TNF-and its receptors and causes lysis of the cells that produce TNF- . Srinivasan et al used infliximab and daclizumab in combination therapy for patients who developed SR GvHD after non myeloablative HSCT in adult patients. All 12 patients treated with the combination therapy had complete resolution of GvHD in all involved organs. The Kaplan-Meier probability of survival was 100% at 100 days and 73% at 200 days after transplantation. Rao et al in their study used the same regimen (infliximab and daclizumab) in pediatric population who underwent HSCT for immunodeficiency. In their study 86% (19/22) patients responded with a median response time of 15 days after start of monoclonal antibody therapy. 12/22 (54%) had CR, and 7/22 (32%) had a PR while 3 patients had no response to treatment. At a median follow-up of 31 months 68% of the patients were alive.

As of Jan 2010 Daclizumab is not available due to manufacturer related issues. Basiliximab is another chimeric murine-human IL-2 receptor antagonist, with a half-life of around 7 days. It's mechanism of action is similar to daclizumab and it has been used in SR GVHD as monotherapy. Massenkeil et al in their study of 17 patients with steroid refractory GvHD showed the 53% of patients had a complete response, 18% had a partial response and 29% had no response. Recently Funke et al in their study of 34 patients with SR GvHD, showed a CR rate of 84% for skin, 48% of gut and 26% of patients with liver GvHD. However it is difficult to compare one study with another due to lack of uniformity in response definitions, dosing schedules and the number of doses used.

The higher CR rates and survival in the studies by Srinivasan and Rao et al were possibly due to the following factors:

1. Use of combination therapy of monoclonal antibodies, selectively inhibiting alloreactive T cells by targeting 2 different cytokines involved in the pathophysiology of GvHD;
2. Rapid taper of steroids, thereby decreasing the steroid induced side effects like infections;
3. Prophylactic use of antimicrobials (antibiotics and antifungals) and close monitoring for viral reactivation.

These factors led to decrease in infection related morbidity and mortality in this population of heavily immunosuppressed patients; thus contributing to the improved survival in these studies.

Overall CR rates for SR GvHD have ranged from 9% to 54% with a median of 26%. Mostly these results are based on single center experience, with small sample sizes, and these studies are not comparable. There is no standard of care; however infliximab may be used as monotherapy if a diagnosis of SR GvHD has been made. The only promising treatment with infliximab and daclizumab is not possible to give now due to unavailability of daclizumab from January 2010. Basiliximab has not been used in combination therapy with other monoclonal antibodies. Combination therapy with infliximab and basiliximab will target two different points in the cytokine cascade and selectively control proliferation of activated T cells. As this combination has not been used before it is difficult to predict the safety and efficacy profile.

ELIGIBILITY:
Inclusion Criteria:

* Any patient with either progressive aGvHD or Steroid Refractory aGvHD after Bone marrow transplant
* Prophylactic GvHD therapy with cyclosporine, tacrolimus, MMF, or sirolimus can be continued.
* Patients with late onset acute GvHD will be eligible
* Patients should have an absolute neutrophil count (ANC) of >500µL
* Patients with renal dysfunction or veno-occlusive disease are eligible

Exclusion Criteria:

* Patient should not be getting any other experimental therapy for aGvHD
* Patients with active uncontrolled life threatening infection (s) from viral, bacterial, fungal or other organisms will be excluded. Patients with HIV infection will be excluded
* Patients who are pregnant, breast feeding, or if sexually active and unwilling to use effective birth control for the duration of this study will be excluded
* Patients with NYHA Class III or IV heart failure will be excluded

Ages: 6 Months to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2011-12; Primary Completion 2015-12 (Actual); Study Completion 2016-09-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rajinder S Bajwa, MD, Principal Investigator — Nationwide Children's Hospital
Locations (3):
- United States (3):
  - University of Florida College of Medicine, Gainesville, Florida
  - Nationwide Children's Hospital, Columbus, Ohio
  - Methodist Healthcare System of San Antonio, San Antonio, Texas

REFERENCES:
- [Background] Srinivasan R, Chakrabarti S, Walsh T, Igarashi T, Takahashi Y, Kleiner D, Donohue T, Shalabi R, Carvallo C, Barrett AJ, Geller N, Childs R. Improved survival in steroid-refractory acute graft versus host disease after non-myeloablative allogeneic transplantation using a daclizumab-based strategy with comprehensive infection prophylaxis. Br J Haematol. 2004 Mar;124(6):777-86. doi: 10.1111/j.1365-2141.2004.04856.x. PMID 15009066
- [Background] Rao K, Rao A, Karlsson H, Jagani M, Veys P, Amrolia PJ. Improved survival and preserved antiviral responses after combination therapy with daclizumab and infliximab in steroid-refractory graft-versus-host disease. J Pediatr Hematol Oncol. 2009 Jun;31(6):456-61. doi: 10.1097/MPH.0b013e31819daf60. PMID 19648797

RESULTS

PARTICIPANT FLOW:
Groups:
- Infliximab and Basiliximab: Other Names:
  Simulect Remicade Monoclonal antibody
  Participants in this research study will receive combination therapy (2 drugs: Infliximab and Basiliximab)once a week for four weeks. Both drugs will be given through the participant's broviac, port or through a vein in the arm. It will take about 4-5 hours to complete the 2-drug combination therapy each week. Participants will be given pre-medications to help prevent reactions to the study drugs.
  Infliximab will be given at a dose of 10mg per Kg per dose. Basiliximab will be given in 10mg doses to patients who weigh less than 35kg. Patients who weigh weigh more than 35kg will receive 20mg doses. Patients will receive both drugs weekly on days 1,8,15 and 22. Each drug will be given 4 times.
  Infliximab and Basiliximab: Participants in this research study will receive combination therapy (2 drugs: Infliximab and Basiliximab)once a week for four weeks.
Period: Overall Study
Arm/Group | Infliximab and Basiliximab
Started | 11
Completed | 11
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Infliximab and Basiliximab
Number analyzed (Participants) | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 8
  Between 18 and 65 years | 3
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 8

OUTCOME MEASURES:

1. Primary Outcome: Complete Response Rate Determination
Description: Complete response was defined as complete resolution of all signs and symptoms of GvHD in all organs using the Modified Glucksberg grading of acute graft versus host disease scale. The score used for GvHD grading complete response was "0" in all evaluable organs.
Time Frame: 28 days
Population: The study was closed prematurely as the study sponsor could not supply the medication any further. The study had not enrolled enough subjects to do a valid statistical analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Infliximab and Basiliximab
Number analyzed (Participants) | 10
Participants | 10

ADVERSE EVENTS:
Arm/Group | Infliximab and Basiliximab
Serious Adverse Events (participants affected / at risk) | 1/11
Other Adverse Events (participants affected / at risk) | 0/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Infliximab and Basiliximab (N=11)
ALT (Hepatobiliary disorders) | 1 (1) — increased ALT

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No